CLINICAL TRIAL: NCT07204847
Title: Prognostic Impact of Guideline-recommended Timing for Invasive Strategy in NSTEMI: a Prospective Real-world Study
Brief Title: Prognostic Impact of Guideline-recommended Timing for Invasive Strategy in NSTEMI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Nīmes (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-12-185
Record Dates: First submitted 2025-09-15; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: NSTEMI; NSTE-ACS (NSTEMI and UA); NSTEMI - Non-ST-Segment Elevation Myocardial Infarction
Keywords: NSTEMI; NSTE-ACS; Invasive strategy timing; Early or delayed intervention
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early intervention: Invasive coronary angiography within 24 hours after diagnosis
- Delayed intervention: Invasive coronary angiography more than 24 hours after diagnosis

SUMMARY:
The objective of this multicentric observational study is to evaluate the prognostic influence of adherence or non-adherence to the recommended coronary angiography timeframe (within 24 hours) and the six-month prognosis of the patients.

DETAILED DESCRIPTION:
Primary Objective: To describe the predictive values (sensitivity and specificity) of the timing of coronary angiography after the diagnosis of NSTEMI.

Secondary Objective: To evaluate an optimal threshold for the timing of coronary angiography that predicts poor prognosis at 6 months (Composite MACCE criterion including all-cause death, recurrent myocardial infarction, hospitalization for cardiac reasons, stroke) (MACCE = Major Adverse Cardiac and Cerebral Events, stroke = cerebrovascular accident).

Comparisons:

Comparison of severe events at 6 months (Composite MACCE criterion including all-cause death, recurrent myocardial infarction, hospitalization for cardiac reasons, stroke) based on the timing of coronary angiography after the diagnosis of NSTEMI according to recommendations (within 24 hours vs. more than 24 hours).

Comparison of severe events at 6 months (all-cause death, recurrent myocardial infarction, hospitalization for cardiac reasons, stroke, considered separately) based on the timing of coronary angiography after the diagnosis of NSTEMI according to recommendations (within 24 hours vs. more than 24 hours).

Comparison of severe events at 1 month (Composite MACCE criterion including all-cause death, recurrent myocardial infarction, hospitalization for cardiac reasons, stroke) based on the timing of coronary angiography after the diagnosis of NSTEMI according to recommendations (within 24 hours vs. more than 24 hours).

Comparison of the occurrence of severe events (Composite MACCE criterion including all-cause death, recurrent myocardial infarction, hospitalization for cardiac reasons, stroke, treated as survival data) based on the timing of coronary angiography after the diagnosis of NSTEMI according to recommendations (within 24 hours vs. more than 24 hours).

Additional Descriptions:

Description of the prevalence of patients for whom the recommended timing of coronary angiography is followed.

Comparison of the characteristics of patients who underwent coronary angiography within 24 hours versus those who did not (age, LVEF (left ventricular ejection fraction), troponin level, creatinine, NYHA class (New York Heart Association heart failure classification)).

Comparison of the length of hospitalization based on the timing of coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chest pain with or without ECG changes
* Elevation of troponin level > 90th percentile or a significant increase between two dosages
* Significant or non-significant coronary lesion confirming the diagnosis of coronary artery disease on coronary angiography (coronary angiography mandatory before inclusion to confirm NSTEMI)

Exclusion Criteria:

* STEMI (ST-segment elevation myocardial infarction) or equivalent (defined as chest pain with ECG changes and troponin elevation > 5 times the normal with an occluded artery (TIMI 0, 1, or 2) during initial coronary angiography)
* Very high-risk NSTEMI (hemodynamic instability, cardiogenic shock, recurrent/refractory chest pain despite optimal medical treatment, life-threatening arrhythmia, mechanical complication, heart failure clearly related to NSTEMI, ST depression > 1mm/6 leads with ST elevation in aVR and/or V1) for which urgent coronary angiography is mandatory
* Unstable angina (acute coronary syndrome without troponin elevation)
* Troponin elevation without chest pain or symptoms suggestive of NSTEMI
* Recovered cardiac arrest
* Contraindication to coronary revascularization or coronary angiography
* Other diagnoses considered after coronary angiography (e.g., myocarditis, Takotsubo syndrome)
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The included patients are those diagnosed with NSTEMI who have undergone coronary angiography as recommended, with no changes to the subsequent patient follow-up
Sampling Method: Non-Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Describe the predictive value of the timing of invasive coronary angiography on a composite criteria of overall mortality, recurrent myocardial infarction, stroke, hospitalization for heart failure at 6 months | From enrollment to 6 months
  Sensibility and specificity, positive and negative predictive values

SECONDARY OUTCOMES:
Evaluation of the optimal timing of invasive coronary angiography predicting a negative outcome at 6 months | From enrollment to 6 months
  Using a receiver operating characteristic (ROC) curve
Comparison of the composite criteria of an invasive coronary angiography within 24h and after 24h at 6 months | From enrollment to 6 months
  Composite of overall mortality, recurrent myocardial infarction, stroke and hospitalization for heart failure
Comparison of the composite criteria of an invasive coronary angiography within 24h and after 24h at 1 month | From enrollment to 1 month
  Composite criteria of overall mortality, recurrent myocardial infarction, stroke and hospitalization for heart failure
Comparison of each element of the composite criteria individually at 6 months of an invasive coronary angiography within 24h and after 24h | From enrollment to 6 months
  Overall mortality, recurrent myocardial infarction, stroke and hospitalization for heart failure
Describe the prevalence of patients receiving an invasive in respect to the timing of the guidelines | At enrollment
  Within 24 hours
Comparison of major bleeding at 6 months | From enrollment to 6 months
Length of in-patient stay | 6 months
  Duration in days between the date of admission at the participating hospital and the date of discharge during the index hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fox KA, Clayton TC, Damman P, Pocock SJ, de Winter RJ, Tijssen JG, Lagerqvist B, Wallentin L; FIR Collaboration. Long-term outcome of a routine versus selective invasive strategy in patients with non-ST-segment elevation acute coronary syndrome a meta-analysis of individual patient data. J Am Coll Cardiol. 2010 Jun 1;55(22):2435-45. doi: 10.1016/j.jacc.2010.03.007. Epub 2010 Mar 30. PMID 20359842
- [Background] Mehta SR, Granger CB, Boden WE, Steg PG, Bassand JP, Faxon DP, Afzal R, Chrolavicius S, Jolly SS, Widimsky P, Avezum A, Rupprecht HJ, Zhu J, Col J, Natarajan MK, Horsman C, Fox KA, Yusuf S; TIMACS Investigators. Early versus delayed invasive intervention in acute coronary syndromes. N Engl J Med. 2009 May 21;360(21):2165-75. doi: 10.1056/NEJMoa0807986. PMID 19458363
- [Background] Kofoed KF, Kelbaek H, Hansen PR, Torp-Pedersen C, Hofsten D, Klovgaard L, Holmvang L, Helqvist S, Jorgensen E, Galatius S, Pedersen F, Bang L, Saunamaki K, Clemmensen P, Linde JJ, Heitmann M, Wendelboe Nielsen O, Raymond IE, Kristiansen OP, Svendsen IH, Bech J, Dominguez Vall-Lamora MH, Kragelund C, Hansen TF, Dahlgaard Hove J, Jorgensen T, Fornitz GG, Steffensen R, Jurlander B, Abdulla J, Lyngbaek S, Elming H, Therkelsen SK, Abildgaard U, Jensen JS, Gislason G, Kober LV, Engstrom T. Early Versus Standard Care Invasive Examination and Treatment of Patients With Non-ST-Segment Elevation Acute Coronary Syndrome. Circulation. 2018 Dec 11;138(24):2741-2750. doi: 10.1161/CIRCULATIONAHA.118.037152. PMID 30565996
- [Background] Kite TA, Kurmani SA, Bountziouka V, Cooper NJ, Lock ST, Gale CP, Flather M, Curzen N, Banning AP, McCann GP, Ladwiniec A. Timing of invasive strategy in non-ST-elevation acute coronary syndrome: a meta-analysis of randomized controlled trials. Eur Heart J. 2022 Sep 1;43(33):3148-3161. doi: 10.1093/eurheartj/ehac213. PMID 35514079